CLINICAL TRIAL: NCT06179147
Title: Effect of Cervical Traction on Oxytocin Level and Postpartum Hemorrhage
Brief Title: Cervical Traction and Postpartum Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, İlkay Ünal, associate professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ILKAYUNAL-DOKTORATEZI-2023
Record Dates: First submitted 2023-09-08; First posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Postpartum Hemorrhage
Keywords: Postpartum hemorrhage; oxytocin; cervical traction
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Intervention Model Description: There are two groups: the cervical traction group (intervention group) and the control group.
Who Masked: Participant
Masking Description: Simple Random Numbers Table was used as the randomization method for sample selection. In this method; Randomly sorted algorithm was created at the maximum allowed percentage and 10% deviation in total 100 samples. In the algorithm, 100 sample (female) groups for both groups; Up to 200 randomly sorted as A and B. Intervention group: A, Control group: B. The sample taken according to the order in the list on the data collection days; It was accepted as group A or B (Piantdosi S, 2005; Pocock SJ, 1983; Rosenberger WF, 2002). The primary outcome measure of the RCT study was the difference between the cervical traction group and the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cervical traction group (intervention group) (Experimental): Immediately after the placenta was expelled, clamping with collum overpens and controlled traction visible through the vaginal introitus were applied to the women in the intervention group of the study. Traction was applied for 90 seconds.
  Interventions: Other: cervical traction
- control group (No Intervention): No procedure was applied to the women in the control group after the placenta was expelled.

INTERVENTIONS:
Other: cervical traction — Traction of the uterine cervix applied in the study; It is the process of pulling the anterior and posterior lips of the cervix towards the intraoitus, downwards and backwards for approximately 90 seconds using overpens. Traction is applied until the cervix reaches the level of vaginal introitus. It is a cost-effective, new, simple intervention with no reported adverse effects.
  Arms: cervical traction group (intervention group)

SUMMARY:
The purpose of the research conducted within the scope of the doctoral thesis study is to evaluate the effect of cervical traction applied at the end of the third stage of childbirth on the oxytocin level and postpartum bleeding (hemoglobin level, estimated blood loss, and amount of bleeding measured with a bleeding tracking bag). The study included 100 women in the intervention group and 100 women in the control group, all of whom met the inclusion criteria. Data were collected throughout the research via an Introduction Information Form, Hemoglobin and Hematocrit Measurement, Calculation of Estimated Blood Loss (modified formula of Gross (1983)), Oxytocin Measurement, and Measurement of bleeding amount with the Bleeding Tracking Bag. Blood was drawn twice from all participating women. The hemoglobin levels of the women were determined with these collected blood samples, and the change before and after the application was identified. Additionally, the oxytocin hormone in the blood was also examined. The change in oxytocin hormone levels before and after application, the difference between groups, and the change within the women themselves were identified. Besides this, the Bleeding Tracking Bag was placed under the women after the birth of the fetus and the amount of bleeding was measured. The Bleeding Tracking Bag was placed under the woman after the placenta was expelled, left for 15 minutes, and the amount of blood accumulated in the bag was recorded in "ml". "Hemoglobin and Hematocrit measurement" was performed when the woman was in the obstetrics ward, when cervical dilatation was 10 cm, and at the end of the 6th hour after birth. Blood taken into the purple cap EDTA tube was delivered daily to an external special laboratory. For determining the "oxytocin" level, 5 ml of blood was taken into the gel blood collection tube when cervical dilatation was 10 cm. After placing the bleeding tracking bag under the woman, cervical traction was applied to the intervention group for 90 seconds. To determine the effect on the oxytocin level after 15 minutes (990 seconds) of applying traction, a second 5 ml blood was taken into the gel blood collection tube. The blood taken was centrifuged by the researcher (PhD student) for 10 minutes and separated into its serum. The separated serums were pipetted into a 1.5 ml Eppendorf tube and stored at -80°C after labeling the tubes.

DETAILED DESCRIPTION:
The research is a randomized controlled intervention study planned to evaluate the effect of the cervical traction maneuver applied at the end of the third stage of labor on oxytocin level and postpartum bleeding. The population of the research consisted of women who gave birth vaginally in the hospital where the research will be conducted during the research (1100 vaginal births between November 2022 and May 2023). realized). The sample of the study consisted of 202 women who gave birth vaginally, where vacuum and forceps were not used, in a training and research hospital obstetrics clinic in Turkey, who met the sample selection criteria and agreed to participate in the study (Intervention group: 102 women; Control group: 100 women). Two women in the intervention group were excluded from the study due to the diagnosis of placenta acreata. The study was completed with 200 women. The smallest sample size to be taken; In order to find the significant difference between the groups, repeated measure analysis of variance (ANOVA) was determined by performing Power (Gpower) analysis under the test. Because, in the study, three different variables will be measured in order to determine the oxytocin level, hemoglobin and hematocrit level, and the amount of bleeding with the bleeding follow-up bag. In the analysis, 196 cases were found sufficient by taking α=0.05 and f=0.25 with 80% power. The sample size was taken as 200 cases against the possibility of data loss.

Simple Random Numbers Table was used as the randomization method for sample selection. In this method; Randomly sorted algorithm was created at the maximum allowed percentage and 10% deviation in total 100 samples. In the algorithm, 100 sample (female) groups for both groups; Up to 200 randomly sorted as A and B. Intervention group: A, Control group: B. The sample taken according to the order in the list on the data collection days; It was accepted as group A or B (Piantdosi S, 2005; Pocock SJ, 1983; Rosenberger WF, 2002). The primary outcome measure of the RCT study was the difference between the cervical traction group and the control group.

Dependent variables of the research; Oxytocin level, hematocrit and hemoglobin value and amount of bleeding are the independent variables; It is the application of cervical traction.

Data were collected using the Introductory Information Form, the formula for Calculated Blood Loss (Gross's modified formula), measuring the oxytocin level and determining the amount of bleeding using Brass-V Drape (bleeding monitoring bag).

1. Introductory Information form:

   The Introductory Information Form, created as a result of the literature review, consists of three sections: Socio-demographic Characteristics, Obstetric Characteristics and Characteristics of the Birth and Postpartum Period. There are a total of 25 questions in the Introductory Information Form (Erkaya R, 2019; Küçükoğlu S, 2019; Hamdy A, et al, 2019; Hamdy A, 2015; Gross JB, 1983).
2. Hemoglobin and Hematocrit Measurement:

   Hemoglobin and hematocrit measurements were taken in all women in the intervention and control groups in the second stage of labor, when cervical dilatation was 10 cm and at the sixth hour after the birth of the fetus. This measurement was performed twice throughout the entire study. For measurement, 2 ml of whole blood was taken into a purple-capped EDTA tube from the vascular access (with branule) opened during the admission of the pregnant women to the delivery room, and the tube was mixed by slowly turning it upside down 5-6 times as soon as the blood was taken to prevent clots from forming in the tubes. Evaluation of hemoglobin and hematocrit was performed with the purchase of services from a private laboratory outside the hospital. The blood taken was delivered to the laboratory where the measurement would be made within seven hours.
3. Calculation of Estimated Blood Loss:

   The amount of blood loss in women was calculated by the researcher using Gross (1983)'s modified formula (Estimated Blood Volume (EBV), estimated blood volume (mL) calculated as weight in kg x 85). For the formula, the Estimated Blood Volume (TKH) was determined first. After calculating THR with the formula "kgx85", Calculated Blood Loss (HKK) was obtained by multiplying the difference between THR and prenatal and postnatal hematocrit values by the average of prenatal and postnatal hematocrit values (Gross JB, 1983).
4. Oxytocin measurement:

   When cervical dilatation is 10 cm and 990 sec after placenta separation. Blood was taken for measurement twice. The reason why cervical dilatation is evaluated when it is 10 cm; According to Roberts and Wolley (1996), the Ferguson reflex is generally activated when the presenting part of the fetus reaches at least +1 level (past the descending ischial spines). At this point, involuntary straining pressure occurs. Hamdy (2015) stated that the mechanism of action of the cervical traction maneuver can be explained by the Ferguson reflex. For this reason, oxytocin level was measured in the second phase before the intervention.

   The second blood draw for oxytocin measurement is; It was performed at 990 sec (16 min. 30 sec) after delivery of the placenta. Oxytocin measurement was carried out by purchasing service from a private laboratory, as it was not a routine evaluation in the hospital where the research data would be collected. While taking blood, vascular access was used for pregnant women during their hospitalization in the delivery room. In case of giving parenteral fluid to the pregnant during labor, a separate vascular access was used for the blood to be taken from the pregnant.
5. Measurement of the amount of bleeding:

A Brass-V Drape (bleeding monitoring bag) was placed under the woman's hip to calculate the amount of bleeding after the placenta came out at the end of the third stage of labor. The bag was kept under the woman until oxytocin measurement (990 sec=16 min. 30 sec).

The research process was carried out in seven steps. The researcher did not make any application to the pregnant women during labor, the routine application and follow-up of the women were done by the midwives and physicians in the clinic. The researcher identified the women and took blood samples. Additionally, cervical traction was applied under the supervision of the responsible physician. The amount of bleeding was determined by the researcher using the Brass V Drape (Bleeding Bag). The women who underwent cervical traction formed the Intervention group (A), and the women who were routinely applied in the clinic without intervention constituted the Control group (B). Groups of women were determined with a table of random numbers.

In addition, in case of parenteral fluid administration to the woman during labor, a separate vascular access was used for the blood taken from the woman.

For intervention group (A):

* First step: An Introductory Information Form was applied to all women who agreed to participate in the study.
* Second step: In the second stage of labor, when cervical dilatation was 10 cm, blood was drawn from the vascular access opened during their admission to the delivery room to evaluate hemoglobin, hematocrit and oxytocin levels. This measurement was used to calculate blood loss as a prenatal measurement. The reason for oxytocin measurement is; According to Roberts and Wolley (1996), the Ferguson reflex is generally activated when the presenting part of the fetus reaches at least +1 level (past the descending ischial spines). At this point, involuntary straining pressure occurs. Hamdy (2015) stated that the mechanism of action of the maneuver he described can be explained by the Ferguson reflex. For this reason, the oxytocin level before the intervention was measured in the second phase.
* Third step: After the placenta came out (at the end of the third stage of labor), the researcher, paying attention to aseptic techniques, placed a Brass-V Drape (bleeding monitoring bag) under the woman's hip to calculate the amount of bleeding. The bag was kept under the woman until oxytocin measurement (990 sec=16 min. 30 sec).
* Fourth step: Following the birth of the placenta, women in the intervention group were subjected to continuous downward and backward traction on the anterior and posterior lips of the cervix with overpens for 90 seconds. Traction was performed until the cervix reached the vaginal introitus level. This process was applied by the researcher. During traction application with overpens, maneuvers were made in accordance with aseptic technique.
* Fifth step: The oxytocin level of the women in the intervention group was measured 990 seconds after the placenta came out. For oxytocin measurement, blood was taken from the vascular access opened during admission to the delivery room. Oxytocin level increases at the 15th minute after birth (Buckley S, 2015). The Bleeding Monitoring Bag was lifted from under the woman and the amount of bleeding was measured. Routine care of the fourth stage of labor especially includes monitoring and evaluation of PPH.
* Sixth step: Hemoglobin and hematocrit levels were checked 6 hours after the birth of the fetus. This measurement was used to calculate blood loss as a postpartum measurement.
* Seventh step: The amount of women's blood loss was calculated by the researcher using Gross (1983)'s modified formula (Estimated Blood Volume (EBV), estimated blood volume (mL) calculated as weight in kg x 85).

For the control group (B):

* First step: An Introductory Information Form was applied to all women who agreed to participate in the study.
* Second step: In the second stage of labor, when cervical dilatation was 10 cm, blood was taken from the vascular access opened during admission to the delivery room to evaluate hemoglobin, hematocrit and oxytocin levels. This measurement was used to calculate blood loss as a prenatal measurement. The reason for oxytocin measurement is; According to Roberts and Wolley (1996), the Ferguson reflex is generally activated when the presenting part of the fetus reaches at least +1 level (past the descending ischial spines). At this point, involuntary straining pressure occurs. Hamdy (2015) stated that the mechanism of action of the maneuver he described can be explained by the Ferguson reflex. For this reason, the oxytocin level before the intervention was measured in the second phase.
* Third step: After the placenta came out (at the end of the third stage of labor), the researcher, paying attention to aseptic techniques, placed a Brass-V Drape (bleeding monitoring bag) under the woman's hip to calculate the amount of bleeding after the placenta came out. The bag was kept under the woman until oxytocin measurement (990 sec=16 min. 30 sec).
* Fourth step: In this step, no intervention was made to the women in the control group.
* Fifth step: In this group, oxytocin level was measured 990 seconds after the placenta came out. For oxytocin measurement, blood was taken from the vascular access opened during admission to the delivery room. Oxytocin level increases at the 15th minute after birth (Buckley S, 2015). The Bleeding Monitoring Bag will be removed from under the woman and the amount of bleeding will be measured. Routine care of the fourth stage of labor especially includes monitoring and evaluation of PPH.
* Sixth step: Hemoglobin and hematocrit levels were checked 6 hours after the birth of the fetus. This measurement was used to calculate blood loss as a postpartum measurement.
* Seventh step: The amount of women's blood loss was calculated by the researcher using Gross (1983)'s modified formula (Estimated Blood Volume (EBV), estimated blood volume (mL) calculated as weight in kg x 85).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18 and over who are not of advanced age
* Non-risky pregnancies (pregnant women without systemic disease, without placental problems such as placenta previa, without fetal problems (eg: low birth weight, intrauterine growth retardation, macrosomia, presentation disorders), those without obstetric problems
* Pregnant women who do not have pre-existing maternal hemorrhagic disorders such as factor 8 or 9 deficiency or VonWillebrand disease,
* Pregnant women with hemoglobin level HB <10 mg / dl and without previous C/S)
* Pregnant women with live fetuses
* Pregnant women at term (those who are older than the 37th week of pregnancy and less than the 42nd week of pregnancy)
* Those who can speak Turkish
* Pregnant women who gave consent to participate in the study were included.

Exclusion Criteria:

* It may occur in the first stage of labor; Pregnant women with pathological conditions such as non-progressive labor, abruption of the placenta, rupture, bleeding, cord prolapse, fetal distress, shoulder impingement,
* Pregnant women who have undergone induction of labor (induction with prostaglandin),
* It may occur in the second stage of birth; Pregnant women with pathological conditions such as shoulder insertion, bleeding and prolongation in the second stage, fetal distess, difficult delivery, vacuum and forceps application,
* It may occur in the third stage of birth; bleeding, placental retention, cavity control, third and fourth degree tear, etc. Pregnant women in situations such as

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women who gave birth vaginally were included
Enrollment: 200 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
postpartum hemorrhage (determined by hemoglobin and hematocrit level) | While the first blood from the women was cervical dilatation 10 cm, the second blood was taken at 6 hours postpartum.
  Hemoglobin, hematocrit, calculated blood loss (Gross's modified formula) and the amount of blood accumulated in Brass V Drape and changes in these parameters of the women in the study before birth (when cervical dilatation was 10 cm) and after birth (6th hour after birth) has been examined.
postpartum hemorrhage (Determined with Bleeding Tracking Bag) | After the placenta was expelled, the bleeding monitoring bag was kept under the woman for 15 minutes.
  The amount of blood (ml) accumulated in the Brass V Drape within 15 minutes after the expulsion of the placenta after the third stage of labor.

SECONDARY OUTCOMES:
Oxytocin level (pg/dL) | The first blood was taken when the cervical dilation was 10 cm, and the second blood was taken after 15 minutes in the intervention group and after 16 minutes and 30 seconds in the control group.
  In order to determine the effect of cervical traction on oxytocin level, prenatal oxytocin levels of the intervention and control groups (when cervical dilatation was 10 cm) were compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University Faculty of Health Sciences, Karşiyaka, İ̇zmi̇r, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The ethics committee, from which the research permission was obtained, was given a document stating that the participant data would not be shared in a different place.